CLINICAL TRIAL: NCT06990425
Title: CLOSM Trial: Groin Closure Using Layered Option for Suture Material
Acronym: CLOSM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Francis Caputo, MD, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-149
Record Dates: First submitted 2025-05-22; First posted 2025-05-25 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Vascular Diseases
Keywords: surgical site complication; vascular surgery; wound healing
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Groin closure after vascular intervention with PDS suture (Active Comparator): Vascular intervention access site closed with PDS suture
  Interventions: Procedure: Groin closure with PDS suture
- Groin closure after vascular intervention with Vicryl suture (Active Comparator): Vascular intervention access site closure with Vicryl suture
  Interventions: Procedure: Groin closure suture material

INTERVENTIONS:
Procedure: Groin closure with PDS suture — Closure of the groin will be performed with PDS suture
  Arms: Groin closure after vascular intervention with PDS suture
Procedure: Groin closure suture material — Closure of the groin will be performed with Vicryl suture
  Arms: Groin closure after vascular intervention with Vicryl suture

SUMMARY:
This is a randomized controlled trial comparing groin closure after vascular intervention with Vicryl suture versus PDS (polydioxanone) suture. This will be a single center trail performed at CCF main campus. Patients will be enrolled in a prospective fashion and will be randomized 1:1 to either PDS or Vicryl closure. Patients undergoing bilateral groin exposure will be randomized to receive both closure types to either groin.

DETAILED DESCRIPTION:
Previous research has provided insights into the properties of various suture materials, yet there remains a gap in our understanding of their relative effectiveness in groin closure specifically within the context of vascular surgery. The lack of definitive evidence on whether Vicryl or PDS (polydioxanone) sutures offer superior outcomes necessitates further investigation. This study aims to address this gap by conducting a head-to-head comparison of these sutures, focusing on their impact on postoperative groin complications.

This is a randomized controlled trial comparing groin closure after vascular intervention with Vicryl versus PDS. This will be a single center trail performed at CCF main campus. Patients will be enrolled in a prospective fashion and will be randomized 1:1 to either PDS or Vicryl closure. Patients undergoing bilateral groin exposure will be randomized to receive both closure types to either groin.

The primary objective of this randomized controlled trial (RCT) is to evaluate the effectiveness of Vicryl versus PDS sutures in reducing groin complications following vascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients > 18 years who undergo ELECTIVE vascular surgery that would require groin incisions
* Patients with to undergo ELECTIVE bilateral groin incisions will be matched to receive closure with PDS in one groin and Vicryl in the other groin

Exclusion Criteria:

1. Age 17 or younger
2. Prisoners
3. Pregnant patients
4. Emergent cases
5. Active groin infection prior to intervention
6. History of prior surgical groin access (re-operative groin)
7. Groin closure after extracorporeal membrane oxygenation (ECMO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of groin complication | 30 days and 1 year
  Number of occurrence of the access site complication

CONTACTS AND LOCATIONS:
Overall Officials: Francis Caputo, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No